CLINICAL TRIAL: NCT02195817
Title: Interventional, Open-label Study of 18 mg Selincro® As-needed Use, in the Treatment of Patients With Alcohol Dependence in Primary Care
Brief Title: Study of 18 mg Selincro® As-needed Use, in the Treatment of Patients With Alcohol Dependence in Primary Care
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated due to enrolment challenges
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15892A; 2013-004688-30 (EudraCT Number)
Record Dates: First submitted 2014-07-17; First posted 2014-07-21 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2017-02

CONDITIONS: Alcohol Dependence
MeSH Terms: conditions — Alcoholism | interventions — nalmefene

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Selincro® 18 mg with continuous psychosocial support: Cohort A (Other): Selincro® as-needed; tablets, orally, 12-week Treatment Period in conjunction with continuous psychosocial support
  Interventions: Drug: Selincro® 18 mg with continuous psychosocial support: Cohort A
- Initial psychosocial support: Cohort B (Other): Initial psychosocial support followed by usual care practice, 12-week Observational Period
  Interventions: Other: Initial psychosocial support: Cohort B

INTERVENTIONS:
Drug: Selincro® 18 mg with continuous psychosocial support: Cohort A
  Other Names: nalmefene
  Arms: Selincro® 18 mg with continuous psychosocial support: Cohort A
Other: Initial psychosocial support: Cohort B
  Arms: Initial psychosocial support: Cohort B

SUMMARY:
To determine the reduction in alcohol consumption in patients with alcohol dependence treated with 18 mg Selincro® as-needed use, in conjunction with continuous psychosocial support in primary care

DETAILED DESCRIPTION:
635 patients are planned (total number of patients) with 475 patients treated with Selincro® (Cohort A) and 160 patients not treated with Selincro® (Cohort B) to determine the reduction in alcohol consumption in patients with alcohol dependence.

Cohort A will comprise patients who maintain a high drinking risk level (DRL, defined by World Health Organization (WHO) as >60g alcohol/day for a man or >40g alcohol/day for a woman), or above, in the period between the Screening and Inclusion Visits.

Cohort B will comprise patients who reduce their alcohol consumption in the period between the Screening and Inclusion visits, that is, patients who do not maintain at least a high DRL at the Inclusion Visit (and are therefore not eligible for treatment with nalmefene according to the SmPC).

ELIGIBILITY:
To ensure the study is broadly representative of primary care clinical practice, minimal inclusion and exclusion criteria are imposed with the main exclusion criteria relating to contraindications to the prescription of Selincro® and reflecting the indication wording in the SmPC.

Inclusion Criteria:

* The patient has alcohol dependence diagnosed according to ICD-10.
* The patient has had a high DRL in the 4 weeks preceding the Screening Visit.
* The patient is a man or woman, aged ≥18 years.
* The patient provides a stable address and telephone number.

Exclusion Criteria:

* The patient has one or more contraindications to the prescription of Selincro®:

  * hypersensitivity to the active substance or to any of the excipients
  * taking opioid analgesics
  * current or recent opioid addiction
  * acute symptoms of opioid withdrawal
  * recent use of opioids suspected
  * severe hepatic impairment (Child-Pugh classification)
  * severe renal impairment (eGFR <30 ml/min per 1.73 m2)
  * a recent history of acute alcohol withdrawal syndrome (including hallucinations, seizures, or delirium tremens)
* The patient has had <6 HDDs (defined by the European Medicines Agency as a day with an alcohol consumption >60g for men or >40g for women) in the 4 weeks preceding the Screening Visit.
* The patient has physical alcohol withdrawal symptoms and requires immediate detoxification for which inpatient treatment is required.
* The patient is currently participating or has recently (in the 4 weeks preceding the Screening Visit) participated in a treatment or support programme for alcohol-use disorders, including Alcohol Anonymous, detoxification treatment, and treatment of alcohol withdrawal symptoms, or the patient is already taking nalmefene or has taken nalmefene in the 6 months preceding the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 378 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in the number of Heavy Drinking Days (HDDs) (days/month) | Baseline to Month 3
  Cohort A

SECONDARY OUTCOMES:
Change in Total Alcohol Consumption (TAC) (g/day) | Baseline to Month 3
  Cohort A
Drinking Risk Level response (RSDRL); defined as a downward shift in Drinking Risk Level (DRL); for patients with a very high DRL at baseline, a shift to medium DRL or below; for patients with a high DRL at baseline, a shift to low DRL or below | Baseline to Month 3
  Cohort A
RLDRL response; defined as a downward shift in DRL to low DRL or below | Baseline to Month 3
  Cohort A
Response defined as ≥70% reduction in TAC | Baseline to Month 3
  Cohort A
Response defined as 0 to 4 HDDs (days/month) | Month 3
  Cohort A
Change in Clinical Global Impression - Severity of Illness (CGI-S) score | Baseline to Week 12
  Cohort A
Clinical Global Impression - Global Improvement (CGI-I) | Week 12
  Cohort A
y-glutamyl transferase (y-GT) | Week 12
  Cohort A
Alanine aminotransferase (ALT) | Week 12
  Cohort A
Aspartate aminotransferase (AST) | Week 12
  Cohort A
Change in 36-item Short-form Health Survey version 2 (SF-36) (only for patients in France and the United Kingdom) | Baseline to Week 12
  Cohort A

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (48):
- France (12):
  - FR010, Bécon-les-Granits
  - FR001, Bordeaux
  - FR005, Bordeaux
  - FR009, Cestas
  - FR012, Chauny
  - FR002, Coulounieix-Chamiers
  - FR008, La Teste-de-Buch
  - FR007, Mont-de-Marsan
  - FR011, Narbonne
  - FR003, Targon
  - FR006, Tonneins
  - FR004, Vieux-Boucau-les-Bains
- Germany (11):
  - DE002, Berlin
  - DE005, Berlin
  - DE006, Essen
  - DE003, Jahnsdorf
  - DE004, Jahnsdorf
  - DE011, Mannheim
  - DE009, Nuremberg
  - DE010, Offenbach
  - DE001, Wallerfing
  - DE007, Weilburg
  - DE008, Weinheim
- Spain (13):
  - ES001, Badalona
  - ES010, Badalona
  - ES003, Barcelona
  - ES004, Barcelona
  - ES008, Canet de Mar
  - ES007, el Prat de Llobregat
  - ES006, Hospitalet Del Llobregat
  - ES009, Hospitalet Del Llobregat
  - ES011, Hospitalet Del Llobregat
  - ES002, Mataró
  - ES013, Matar
  - ES012, Sabadell
  - ES005, Tarragona
- United Kingdom (12):
  - GB011, Ballymena
  - GB008, Belfast
  - GB009, Belfast
  - GB004, Cardiff
  - GB005, Cardiff
  - GB001, Coatbridge
  - GB002, Glasgow
  - GB003, Lanarkshire
  - GB006, Swansea
  - GB007, Swansea
  - GB010, Swansea
  - GB106, Swansea

REFERENCES:
- See also: EMA EudraCT Results: 2013-004688-30 — https://www.clinicaltrialsregister.eu/ctr-search/trial/2013-004688-30/results